CLINICAL TRIAL: NCT07355465
Title: The Effect of Salvadora Persica (Miswak) Compared to Fluoridated Toothpaste on Children's Teeth Diagnosed With Molar-Incisor Hypomineralization (MIH): A Randomized Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Heba sabbagh, professor, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 130-10-24
Record Dates: First submitted 2025-11-20; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Molar Incisor Hypomineralisation
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Salvadora Persica (Miswak) (Experimental): Intervention Group:
  Participants in this group will be provided with Salvadora persica (miswak) sticks and receive training on the correct technique for its use. Miswak sticks, uniform in length and width, supplied fresh from Jeddah Central Market, Saudi Arabia, to the subjects in the test group.
  In this group, subjects will be instructed to brush with the miswak using the rolling technique, advised to use it three times a day under a parent's supervision, and shown how to keep it fresh by cutting off the edge of the miswak every day and storing it in the refrigerator at night.
  Interventions: Other: Salvadora persica (miswak)
- Fluoridated Toothpaste Group (Active Comparator): Control Group:
  Participants in this group were instructed to use only fluoridated toothpaste as part of their oral hygiene routine. Oral hygiene instructions will be given for both groups. Modified bass technique for tooth brushing twice daily, 10 seconds per quadrant, with a 1450 ppm fluoride concentration
  Interventions: Device: Fluoridated Toothpaste

INTERVENTIONS:
Other: Salvadora persica (miswak) — Salvadora persica (miswak) has been traditionally used as a natural toothbrush across various cultures for centuries. It contains several biologically active compounds, including fluoride, silica,
  Arms: Salvadora Persica (Miswak)
Device: Fluoridated Toothpaste — Participants will use fluoridated toothpaste (1450 ppm fluoride) three times daily under parental supervision for 9 months to compare its effects with Nano-hydroxyapatite.
  Arms: Fluoridated Toothpaste Group

SUMMARY:
Molar-Incisor Hypo mineralization (MIH) was first described in 2001 as a developmental enamel defect . It is a condition in which the enamel of at least one first primary molar is affected with a qualitative defect causing abnormal translucency appearing as demarcated opacities; The permanent incisors and second primary molars can also be affected . MIH has adverse consequences on the oral health and child's quality of life. It increases the risk of caries, discomfort and teeth sensitivity .

MIH management comprises a variety of treatment options ranging from total caries removal to the polar opposite treatment option of no caries removal and non-invasive methods used to prevent caries progression . Dental caries prediction and prevention are now more important than dental caries diagnosis and treatment. Recently, the reasons for repairing dental cavities have been narrowed, and caries prevention is being used to reduce caries . Salvadora persica, commonly known as Miswak was used as a toothbrush for many years among many countries . It was reported to have a significant effect on oral health and caries prevention .Other studies have found a consistent link between the use of Miswak and a reduction in oral bacteria. However, a comprehensive assessment of using Miswak in the treatment and control of MIH among young children has yet to be conducted.

Therefore, the aim of this clinical trial is to assess the effect of SalvadoraPersica and fluoridated toothpaste on controlling hypersensitivity and preventing caries among children with MIH in primary schools. Additionally, this trial will evaluate the shade of the hypo-mineralized enamel before and after using SalvadoraPersica and fluoridated toothpaste

ELIGIBILITY:
Inclusion Criteria:

* Healthy children with age ranged between 6-12 years old

  * Presence of at least one first permanent molar and incisor diagnosed with MIH.
  * The MIH-affected teeth will have a clinical presentation of white, creamy, yellow, or brown demarcated opacities

Exclusion Criteria:

* Medically compromised children.
* Unwillingness to participate or be randomly assigned to the study groups.
* Receiving treatment for controlling MIH other than fluoride application

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2026-01-29 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
To Assess the effect of Salvadora Persica on the color of MIH-affected teeth compared to brushing with fluoridated toothpaste | Before intervention as a baseline reading (T0), one month (T1), three months later (T2), and six months later (T3)
  The VITA Easyshade® advance spectrophotometer (VITA Zahnfabrik, Bad Sackingen, Germany) will be used to assess the color of MIH-affected permanent incisors and the adjacent sound enamel

SECONDARY OUTCOMES:
the effectiveness of Salvadora Persica on the hypersensitivity of MIH-affected teeth compared to brushing with fluoridated toothpaste | Before intervention as a baseline reading (T0), one month (T1), three months later (T2), and six months later (T3).
  Hypersensitivity can be measured using a visual analog scale (VAS) and the Schiff sensitivity scale to rate patients' pain This scale ranges from zero, representing "No Pain," to 10, representing the "Worst Pain Possible," and is categorized into four levels: mild (1-3), moderate (4-6), severe (7-9), and very severe to worst pain (10). The Schiff Cold Air Sensitivity Scale is a 4-point scale used to assess dentin hypersensitivity. A score of zero indicates no sensitivity, one signifies mild sensitivity without a request to stop the stimulus, two represents moderate sensitivity with a request to stop or visible discomfort, and three indicates severe sensitivity with a request to stop and physical withdrawal.